CLINICAL TRIAL: NCT06049290
Title: A Multicenter, Open-label, Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of LBL-034 in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Phase I/II Clinical Trial of LBL-034 in Patients With Relapsed Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBL-034-CN001
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-05

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LBL-034 (Experimental): LBL-034 for Injection; Initial dose - MTD; Q2W
  Interventions: Drug: LBL-034 for Injection

INTERVENTIONS:
Drug: LBL-034 for Injection — Initial dose - MTD; Q2W; intravenous infusion
  Other Names: LBL-034

SUMMARY:
This is a single-arm, open-label, multicenter, dose-escalation, and dose-expansion phase I/II clinical study to evaluate the safety, tolerability, pharmacokinetics, immunogenicity, and efficacy of LBL-034 in patients with Relapsed/Refractory Multiple Myeloma (R/R MM).

DETAILED DESCRIPTION:
A multicenter, open-label, phase I/II clinical study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of LBL-034 in patients with relapsed/refractory multiple myeloma.

This trial includes two parts: phase I and phase IIa study.

The dose escalation and dose expansion studies for LBL-034 will be conducted in the phase I study to evaluate safety, tolerability and determine RP2D.

The efficacy of LBL-034 in the treatment of R/R MM and R/R leukaemia plasmacytic (plasma cell leukemia, PCL) will be evaluated in Phase IIa study.Phase IIa clinical study will be conducted after obtaining the RP2D.Determine the specific dosing regimen in Phase IIa based on the safety, PK and other data from Phase I clinical studies.Phase IIa clinical study includes 4 cohorts.This trial requires collection of biological samples from all subjects for relevant testing.

This clinical trial will enroll 342 patients in Phase I and Phase IIa studies.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the trial treatment regimen and visit schedule, voluntarily enroll in the study, and sign the written informed consent form;
2. Age ≥ 18 years at the time of signing the informed consent;
3. Eastern Cooperative Oncology Group (ECOG) Performance Status Scale≤ 1；
4. Documentation of initial diagnosis of multiple myeloma according to IMWG diagnostic criteria；
5. Have a life expectancy of at least 12 weeks；
6. Fertile men and women of childbearing age are willing to take effective contraceptive measures (including abstinence, intrauterine devices, hormonal contraception, and correct use of condoms) from the signing of the informed consent form to 6 months after the last dose of the investigational drug; women of childbearing age include premenopausal women and women who had menopause less than two years ago. Blood pregnancy test results must be negative for women of childbearing age within 7 days prior to the initial dose of the investigational drug.

Exclusion Criteria:

1. Subjects who underwent major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to the initial use of the investigational drug,or require elective surgery during the trial period;
2. Use of immunomodulatory drugs within 14 days prior to the initial use of the investigational drug, including but not limited to thymosin, interleukin-2, and interferon；
3. Systemic use of corticosteroids or other immunosuppressants within 14 days prior to the initial use of the investigational drug;The following conditions are excluded: Treatment with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; short-term use of glucocorticoids for preventive therapy (e.g., to prevent contrast allergy);
4. Patients with active hepatitis B or C；
5. Subjects with an active infection that currently requires intravenous anti infective therapy;
6. The patient has a Medical history of immunodeficiency, including HIV antibody positive;
7. Women during pregnancy or lactation;
8. The investigator believes that the subject has other conditions that may affect compliance or are not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy).
  ORR [including the rates of Strin-gent complete response(sCR),complete response (CR) ,Very good partial response(VGPR),and partial response (PR)], evaluated based on the 2016 IMWG criteria(Cohorts 1, 2, and 3) and 2013 IMWG criteria(Cohort 4), refers to the percentage of study subjects who achieve a complete response or partial response. It was used to evaluate the efficacy of LBL-034 in Phase IIa study .
Dose-limiting toxicities（DLT） | The DLT observation period starts from the first dose until 4 weeks after the full dose first administration (including the step-up dosing period, if any).
  DLT describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.DLT is defined as toxicity (possible adverse events related to LBL-034) during the DLT observation period . It was used to evaluate the safety of LBL-034 in Phase I study .
Maximum tolerated dose (MTD) | The MTD observation period starts from the first dose until 4 weeks after the full dose first administration (including the step-up dosing period, if any).
  MTD is defined as the hightest dose level at which no more than 1 out of 6 subjects experiences a DLT during the first cycles. It was used to evaluate the tolerability in Phase I.

SECONDARY OUTCOMES:
Cmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy)
  Maximum drug concentration in plasma after administration.
Tmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy)
  After administration,Time to reach maximum drug concentration in plasma.
Immunogenicity | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy)
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects.Immunogenicity refers to the performance that can elicit an immune response.
Minimal Residual Disease (MRD) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy)
  MRD-negative rate: Refers to the percentage of subjects who achieve MRD negativity at any time point after the initial dose and before disease progression or the initiation of a new anti-tumor therapy.
Duration of Response(DOR） | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy)
  DOR is defined as the duration from earliest date of disease response (CR、PR 、iCR or iPR) until earliest date of disease progression or death from any cause(if occurring sooner than progression).
sBCMA | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy)
  serum B-cell maturation antigen(Detect the change of sBCMA in serum)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, Principal Investigator — Peking University People's Hospital
Locations (26):
- China (26):
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The Afliliated Hospital of Guizhou Medical Univeristy, Guiyang, Guizhou
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - The First Affiliated Hospital of Henan University, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shengyang, Liaoning
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Shanghai Fourth People's Hospital, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University (Xibei Hospital), Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - Institute of hematology & blood diseases hospital, chinese academy of medical sciences & peking union medical college, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No